CLINICAL TRIAL: NCT05929378
Title: A Comparative Study of 3-point With 1-point Mesh Fixation in TAPP Surgery for Patients With Gilbert Type III Inguinal Hernia: A Randomized Controlled Trial
Brief Title: A Comparative Study of 3-point With 1-point Mesh Fixation in TAPP for Gilbert Type III Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Collaborators: Guang'an People's Hospital (Unknown); Pengan County People's Hospital (Other); People's Hospital of Yilong County (Unknown); Nanbu Hospital of County Chinese Medicine (Other); Nanchong Jialing District People's Hospital (Unknown); Langzhong People's Hospital (Unknown); Langzhong Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Principal Investigator, Yunhong Tian, Director of Gastrointestinal, Colorectal and Hernia Surgery, Nanchong Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023031
Record Dates: First submitted 2023-06-17; First posted 2023-07-03 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hernia, Inguinal; Chronic Pain; Seroma; Recurrence; Infections; Hematoma
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain; Seroma; Recurrence; Infections; Hematoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-point fixation group (Experimental): Lightweight Mesh Fixation with 3-point Fixation. First fixation is in cooper ligament. Second fixation is in the back of rectus abdominis. Third fixation is in the later of tractus iliopubicus.
  Interventions: Procedure: Lightweight mesh fixation
- 1-point fixation group (Active Comparator): Lightweight Mesh Fixation with 1-point Fixation in the back of rectus abdominis.
  Interventions: Procedure: Lightweight mesh fixation

INTERVENTIONS:
Procedure: Lightweight mesh fixation — Lightweight mesh fixation in 3 points

SUMMARY:
This study was designed to compare the outcome of 3 point with 1 point lightweight mesh fixation in TAPP surgery for patients with type Ⅲ gilbert inguinal hernia. The main outcome include seroma, chronic pain, recurrence, et al.

ELIGIBILITY:
Inclusion Criteria:

Unilateral indirect inguinal hernia according to preoperative physical examination and imaging examination.

The inclusion criteria were as follows: primary indirect inguinal hernia classified as Gilbert III (defect size diameter ≥3cm, including scrotal hernias)

Exclusion Criteria:

Age below 18 years or older than 80. Direct hernia, femoral hernia, recurrent hernia, incarcerated hernia, strangulated hernia, and other types of hernias.

Patients not suitable for general anesthesia. Patients requiring open surgery; patients requiring emergency surgery Loss to follow-up or communication difficulties, or poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
recurrence | 6 months
  Check for recurrence by clinical examination or ultrasound at 6 months postoperatively
Postoperative pain | 6 months
  The visual analog scale (VAS) was adopted for pain evaluation 2 days, 3 months, and 6 months postoperatively. The scale range from 0 to 10, with 0 meaning no pain and 10 meaning the worst pain.

SECONDARY OUTCOMES:
postoperative complications | 6 months
  Including infection, seroma, hematoma

CONTACTS AND LOCATIONS:
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China